CLINICAL TRIAL: NCT04643769
Title: Phase 1b Double-Blind, Placebo-Controlled, Ascending Dose Trial: ORIN1001 in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Evaluation of Oral ORIN1001 in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Partnership activities ongoing
Sponsor: Orinove, Inc. (Industry)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ORIN1001-002
Record Dates: First submitted 2020-11-11; First posted 2020-11-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo-controlled, double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- 25 mg ORIN1001 (Active) (Experimental): 25 mg ORIN1001
  Interventions: Drug: ORIN1001
- 50 mg ORIN1001 (active) (Experimental): 50 mg ORIN1001
  Interventions: Drug: ORIN1001
- 100 mg ORIN1001 (active) (Experimental): 100 mg ORIN1001
  Interventions: Drug: ORIN1001
- Placebo - 25 mg (Placebo Comparator): Placebo comparator for ORIN1001 at 25 mg
  Interventions: Drug: Placebo
- Placebo - 50 mg (Placebo Comparator): Placebo comparator for ORIN1001 at 50 mg
  Interventions: Drug: Placebo
- Placebo - 100 mg (Placebo Comparator): Placebo comparator for ORIN1001 at 100 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORIN1001 — Oral tablet - ORIN1001
  Arms: 100 mg ORIN1001 (active); 25 mg ORIN1001 (Active); 50 mg ORIN1001 (active)
Drug: Placebo — Oral tablet - placebo
  Arms: Placebo - 100 mg; Placebo - 25 mg; Placebo - 50 mg

SUMMARY:
This Phase 1b trial is a double-blind, placebo-controlled, multiple ascending dose study to evaluate the safety and tolerability of oral ORIN1001 at 25 mg, 50 mg or 100 mg administered daily for up to 28 days in adult subjects with idiopathic pulmonary fibrosis (IPF) alone or in conjunction with local Standard of Care for IPF (pirfenidone or nintedanib).

A maximum of 24 evaluable subjects will be required to complete the study. The study will consist of 3 dose cohorts each enrolling a maximum of 8 subjects randomized either to the active (5 subjects) group or placebo (3 subjects) group. Each subject will receive daily oral doses of ORIN1001 or placebo for 28 days.

The safety and pharmacokinetic profile will be evaluated in this study and will include cardiovascular and pulmonary endpoints.

DETAILED DESCRIPTION:
This Phase 1b trial is a double-blind, placebo-controlled, multiple ascending dose study to evaluate the safety and tolerability of oral ORIN1001 at 25 mg, 50 mg or 100 mg administered daily for up to 28 days in adult subjects with idiopathic pulmonary fibrosis (IPF) alone or in conjunction with local standard of care (SOC) for IPF (i.e., pirfenidone or nintedanib).

Approximately 24 evaluable subjects will be required for this study. Eligible subjects will be followed for safety through the dose-limiting toxicity (DLT) evaluation period, defined as 28 days after the first dose of ORIN1001.

In the absence of intolerable toxicity, doses will be escalated sequentially with 8 evaluable subjects receiving a maximum of 28 days of ORIN1001 in once-daily doses of 25 mg (Cohort 1), 50 mg (Cohort 2), or 100 mg (Cohort 3) versus matched placebo. Subjects will be stratified based on local SOC for IPF, defined as the stable daily dose of pirfenidone or nintedanib (or neither) received for at least 8 weeks prior to signing the Informed Consent Form (ICF). ORIN1001 or matched placebo will be administered daily until Day 28, unacceptable toxicity, withdrawal for another reason or study termination.

Safety Endpoints will be evaluated and will include adverse events (AEs), serious adverse events (SAEs), and changes in clinical laboratory evaluations as compared to baseline. Safety variables include but are not limited to: vital signs (blood pressure [BP], heart rate [HR], respiratory rate [RR]) and temperature; twelve-lead ECG; clinical laboratory tests (hematology, coagulation profile, clinical chemistry, and urinalysis); concomitant medications; physical examination; body weight; and pulmonary function tests (forced vital capacity [FVC], forced expiratory volume [FEV], and diffusion capacity [DLCO]) at baseline, End-of- Treatment and Follow-up Visits.

Pharmacokinetic (PK) Endpoints will be evaluated on Day 1 and Day 28 and blood collection samples will be obtained from each subject. Exploratory serum biomarker endpoints will be evaluated to assess lung fibrosis and inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. 40-80 years of age (inclusive) when signing the Informed Consent.
2. Diagnosis of IPF or likely IPF per 2018 American Thoracic Society and European Respiratory Society (ATS/ERS) criteria:

   * Study Investigator will confirm IPF diagnosis based on Interstitial Lung Disease (ILD) in consultation with relevant experts through a review of the subject's history, high-resolution computerized tomography (HRCT) scan, and lung biopsy (if applicable).
   * A lung biopsy is not required in the setting of a compatible clinical history and usual interstitial pneumonia (UIP) or probable UIP per HRCT.
   * Study Investigators will verify that a diagnosis of IPF and an HRCT were obtained within 7 years prior to signing the ICF.
3. Continued SOC IPF therapy (consisting of pirfenidone [Esbriet®] OR nintedanib [Ofev®] OR neither) is acceptable, provided stable dosing of the drug for at least 8 consecutive weeks immediately prior to signing the ICF.
4. The effect of ORIN1001 on the developing human fetus, if any, is unknown. Therefore, for the duration of study participation:

   * Women who are postmenopausal for < 1 year before the Screening and not otherwise sterile (e.g., due to a surgical procedure) may be considered of child-bearing potential and require a negative pregnancy test prior to study registration. They must agree to (a) use effective contraception (i.e., hormonal or barrier method of birth control when engaged in heterosexual intercourse) or (b) abstinence throughout the study period AND for 4 weeks after final dosing with the IMP.
   * Men who are not otherwise sterile (e.g., due to a surgical procedure) must agree not to donate sperm and use effective contraception (i.e.,hormonal or barrier method of birth control when engaged in heterosexual intercourse) or abstinence throughout the study period AND for at least 16 weeks (due to the sperm life cycle) after final dosing with the IMP.
5. Written informed consent must be given prior to any study-related procedure that is not part of standard medical care, understanding that the subject may withdraw it at any time without prejudice to future treatment.

Exclusion Criteria:

1. Screening lab values that fail to meet the following criteria will render the subject ineligible for study participation:

   * Platelet count <100 × 109/L. Repeat measurements may be performed, but transfusion, in order to meet eligibility criteria, is not allowed.
   * Hemoglobin <12.9 g/dL (men) and <11.9 g/dL (women).
   * Prothrombin time (PT) or partial thromboplastin time (PTT) >1.5 × upper limit of normal; international normalized ratio (INR) >2.
   * Aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >1.5 × upper limit of normal (ULN).
   * Serum glutamic-oxaloacetic transaminase [SGOT] or serum glutamic pyruvic transaminase [SGPT]) >2.0 × ULN.
   * Kidney disease with estimated glomerular filtration rate <60 mL/min).
2. Forced vital capacity (FVC) ≤40% of predicted normal per site pulmonary function lab protocol.
3. Diffusing capacity of the lungs for carbon monoxide (DLCO) ≤30% of predicted normal as calculated according to the site pulmonary function lab protocol.
4. Forced expiratory volume in one second/forced vital capacity (FEV1/FVC) ratio < 0.7.
5. Documented IPF exacerbation within 3 months of signing the ICF (e.g., >5% or 10% change in FVC and DLCO, respectively).
6. Listing for lung transplantation, defined as the assignment of a lung allocation score or acceptance on the waiting list for lung transplantation.
7. Current and/or uncontrolled cardiovascular condition (e.g., clinically significant arrhythmia or hypertension), >Class II heart failure per New York Heart Association criteria, unstable angina, myocardial infarction, coronary syndrome) within 6 months of Screening which, as judged by the Investigator, might put the subject at risk because of participation in the study.
8. Known cirrhotic liver, chronic liver, or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones). Liver cirrhosis with portal hypertension and active liver infection are exclusionary (note: cured hepatitis C is not considered active).
9. Gastrointestinal disease (e.g., active bleeding or ulcers) or procedure that could interfere with oral absorption or tolerance of the IMP, including difficulty swallowing.
10. Diarrhea >Grade 1 (i.e., increase of >4 stools per day OR >1 watery stool per day OR moderate increase in ostomy output compared to baseline) will render a subject ineligible for participation in this study. Anti-diarrheal medication (e.g., loperamide, sold under the brand name Imodium®, among others) is allowed.
11. Active malignancy within the past 12 months or ongoing active cancer treatment (surgery, radiotherapy, chemotherapy or immunotherapy), except for adequately treated Stage 1 cancer, nonmelanoma skin cancer, or in situ cervical cancer. Cancer in complete remission or requiring only maintenance therapy (e.g., tamoxifen for breast cancer) is not considered active.
12. Known bleeding risk due to platelet dysfunction, or inherited or acquired clotting factor deficiency (e.g., von Willebrand disease, hemophilia).
13. Major trauma or surgery including but not limited to operations involving a major organ (e.g., the cranium, chest, abdomen, or pelvic cavity) OR requiring a lengthy recovery period (e.g., arthroplasty) within 3 months of signing the ICF; or expected surgery during the trial period.
14. Central nervous system hemorrhagic event within 12 months of signing ICF; brain arterio-venous malformation (AVM) or moderate-to-severe ischemic stroke within 6 months of signing ICF.
15. Concurrent use of full-dose therapeutic anti-coagulation (e.g., vitamin K antagonist, dabigatran, hirudin, direct factor Xa inhibitors) or high dose anti-platelet therapy. Aspirin <81 mg/day, prophylactic subcutaneous (SC) heparin or SC low-molecular weight heparin for deep vein thrombosis prophylaxis or heparin flush to maintain intravenous catheter patency are allowed.
16. Long-term use of nonsteroidal anti-inflammatory agents, defined as >4 days per week.
17. Receipt of hematopoietic growth factors, blood or blood product transfusion within 1 week of the first dose of IMP.
18. Disqualifying treatments within 60 days or 5 half-lives (whichever is longer) from Randomization include:

    * Systemic corticosteroids (>10 mg prednisone or equivalent).
    * Systemic immunosuppressive therapy.
    * Investigational agent other than study IMP.
19. Recreational drug use (including amphetamines, cocaine, barbiturates, opiates, benzodiazepines, phencyclidine, and cannabinoids) for the duration of study participation.
20. Clinically significant laboratory abnormality, medical or psychological comorbidity, or concurrent medication that could compromise subject safety, data integrity or requirements for study participation, per site Investigator in consultation with the Sponsor.
21. Inability to attend in-person appointments per current clinical site COVID-19 guidelines and restrictions.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Up to 60 days
  measurement of blood pressure
Heart Rate | Up to 60 days
  measurement of heart rate
Respiratory Rate | Up to 60 days
  Measurement of respiratory rate
Body Temperature | Up to 60 days
  Measurement of body temperature
12-lead ECG | Up to 60 days
  Cardiovascular evaluation to determine intervals including QTc interval
Serum Clinical Chemistry analysis | Up to 60 days
  ALT, albumin, ALP, AST, BUN, Ca, Cl, Cholesterol, Creatinine, CK, CA, Elastase, GGT, glucose, HDL, LDH, lipase, LDL, phosphorus, sodium, Total bilirubin, Total protein, Triglycerides, Uric acid, Lipid panel
Whole blood Hematology analysis | Up to 60 dys
  WBC, RBC, Hb, HCT, MCV, MCH, MCHC, Neu, Lymphocytes, EOS, Bas, PLT
Whole blood Coagulation Parameters | Up to 60 days
  PT, APTT, INR
Urinalysis | Up to 60 days
  Bilrubin, glusoe, ketones, leukocytes, nitrite, blood, pH, specific gravity, protein, urobilinogen
Concomitant medications | Up to 60 days
  Evaluation of other medications taken currently with investigative drug
Physical examination | Up to 60 days
  Medical Health examination, medical history, medicine history, reproductive history, baseline information
Body weight | Up to 60 days
  Body weight in kg
Spirometry | Up to 60 days
  Pulmonary Function Tests: Forced vital capacity (FVC), Forced expiratory volume (FEV)
Height | Up to 60 days
  Height in cm
Body mass index (BMI) | Up to 60 days
  Calculation of BMI using weight (kg) and height (cm)
DLCO - Assessment of diffusion capacity | Up to 60 days
  Lung test to assess diffusion capacity

SECONDARY OUTCOMES:
Blood collection to measure drug concentration over time | Up to 29 days
  Blood collection for evaluation of ORIN1001 exposure. Measurements will assess half life, exposure, maximum concentration, time to maximum concentration and accumulation ratios

OTHER OUTCOMES:
Exploratory biomarkers to evaluate lung fibrosis | Up to 60 days
  Blood collection for evaluation of disease biomarker of lung fibrosis: SP-D, MMP-7 and KL6. Specific biomarker to be determined
Quality of Life Questionnaire | Up to 60 days
  Questionnaire to assess the quality of life during the study period
Exploratory biomarkers to evaluate inflammation | Up to 60 days
  Blood collection for evaluation of inflammation such as cytokines TGF-B and/or IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Frank Averill, MD, Principal Investigator — Sleep, Allergy and Lung Institute
Locations (11):
- United States (11):
  - St. Francis Sleep, Allergy & Lung Institute, Clearwater, Florida
  - Mayo Clinic Hospital, Jacksonville, Florida
  - Avanza Medical Research, Pensacola, Florida
  - Coastal Pulmonary and Critical Care, St. Petersburg, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospital, Iowa City, Iowa
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - Hannibal Clinic, Hannibal, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Duke University Hospital, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No